CLINICAL TRIAL: NCT05171556
Title: IN-USE TOLERANCE STUDY UNDER DERMATOLOGICAL AND OPHTHALMOLOGICAL CONTROLS AND EFFICACY ASSESSMENT
Brief Title: IN-USE TOLERANCE STUDY UNDER DERMATOLOGICAL AND OPHTHALMOLOGICAL CONTROLS AND EFFICACY ASSESSMENT (Face Balm)
Status: Completed | Type: Observational
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Other Study IDs: RV4942A20200169
Record Dates: First submitted 2021-12-10; First posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Hypersensitive; Reactive and Intolerant Skin; Redness-prone Skin; Stinger Subjects
Keywords: Hypersensitive skin; Discomfort sensations; Asian skin; Sensitivity reduction
MeSH Terms: conditions — Hypersensitivity | interventions — Cosmetics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RV4942A arm: RV4942A study product is applied twice a day (morning and evening) on the face, neck and eye contour during the whole study.
  Interventions: Other: Cosmetic product

INTERVENTIONS:
Other: Cosmetic product — RV4942A is a face balm product

SUMMARY:
The aim of this study is to assess the dermatological and ophthalmological tolerance of the investigational product Baume visage / Face balm RV4942A - RY1985 after 21 days of twice daily use on the study areas, under normal conditions of use.

The aim of this study is also to:

* evaluate the cutaneous sensitivity by a stinging test at D1 T0 and D22.
* evaluate the cutaneous sensitivity by a sensitive scale at D1 T0, D1 Timm*, D8 and D22.
* evaluate the soothing efficacy by an efficacy questionnaire at D1 Timm*, D8 and D22.
* evaluate the cosmetic acceptability by a questionnaire at D22.

This study is conducted as a national, monocentric, non-randomized open trial. The 33 subjects in this study (31 subjects on D22) present hypersensitive, reactive and intolerant skin on face. They are stinger subjects, with a dry to very dry skin.

Timm*: 10 to 30 minutes after first application

DETAILED DESCRIPTION:
his study is a national, monocentric, non-randomized open trial, conducted in adults presenting hypersensitive, reactive and intolerant skin on the face, with a dry to very dry skin.

The study includes 3 visits, including subjects' selection:

* V1: Baseline inclusion
* V2: 1 week, intermediate visit
* V3: 3 weeks, study end

The maximal study duration is 25 days.

The evaluation is at 3 times: D1 baseline, D8 at 1 week and D22 at 3 weeks of application of RV4942A - RY1985 with comparison of each time versus baseline.

There are twice-daily applications (morning and evening) of the test product on the face.

ELIGIBILITY:
Inclusion Criteria:

1. Criteria related to the population:

   * Male or Female aged between 18 and 65 years included
   * Asian population (Chinese origin)
   * Dry to very dry skin on the face
   * Subject with phototype I to IV included
   * Subject having signed his/her written informed consent for his/her participation in the study
   * Subject who is currently not participating in another clinical study
   * Subject affiliated to a social security system or health insurance, or is a beneficiary
   * For woman of childbearing potential: use of an effective method of contraception and using it during the whole duration of the study
2. Criteria related to diseases and general health:

   * Stinger subjects (evaluated by a stinger test)
   * Subject with hypersensitive, reactive and intolerant skin on face
   * Subject having a score superior to 4 on a sensitive scale for tightness parameter on the face
   * Subject having a score superior to 4 on a sensitive scale for general discomfort parameter on the face

Exclusion Criteria:

1. Criteria related to the population:

   * For woman of childbearing potential: subject pregnant or breastfeeding or planning to be pregnant during the study
   * Having a dermatological condition liable to interfere with the study data or considered by the Investigator hazardous for the subject or incompatible with the study requirements
   * Having an ophthalmological condition liable to interfere with the study data or considered by the Investigator hazardous for the subject or incompatible with the study requirements
   * Having personal medical history liable to interfere with the study data for the subject or incompatible with the study requirements
   * Having history of abnormal reactions from exposure to sunlight
   * Having taken any previous treatment considered by the Investigator liable to interfere with the study data or incompatible with the study requirements
   * Being under any treatment considered by the Investigator liable to interfere with the study data or incompatible with the study requirements
   * Subject who is not likely to be compliant with study-related requirements
   * Subject deprived of freedom by administrative or legal decision or under guardianship
2. Criteria related to investigational product application areas:

   * Having had any surgery, chemical or significant invasive dermotreatment on the experimental area considered by the Investigator liable to interfere with the study data, before the inclusion visit or foreseeing it for the duration of the study
   * Having applied a skincare or make up product on the study areas the day of the inclusion visit. The usual cleanser is allowed
   * Having received, on the study areas, artificial UV exposure or excessive exposure to natural sunlight within the 2 weeks before the inclusion visit (at Investigator's opinion)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects have been recruited from the panel of the centre. An investigator made a dermatological examination of the subjects before inscription in the panel. Data from this clinical examination, stored in the computer database with the consent of the subjects, can ensure the recruitment; computer software being questioned based on the eligibility criteria of the study.
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2021-05-11 (Actual)

PRIMARY OUTCOMES:
Global tolerance assessment of the investigational product by dermatological evaluation | Change from baseline to just after application and to 3 weeks later
  Dermatological evaluation based on physical and functional signs assessment by the dermatologist
Global tolerance assessment of the investigational product by ophthalmological evaluation | Change from baseline to just after application and to 3 weeks later
  Ophthalmological evaluation based on physical and functional signs assessment by the ophthalmologist

SECONDARY OUTCOMES:
Cutaneous sensitivity by stinging test | Change from baseline to 3 weeks later
  Stinging test is an in vivo methodology that evaluates sensitive skin and consists in application of 10% lactic acid on one nasolabial fold of subject's nasogenian folds
Cutaneous sensitivity by sensitivity scale questionnaire | Change from baseline to 1 week and to 3 weeks later
  Subjects assess the degree of their overall face skin irritation using an Analogue Visual Scale and fill out the sensitivity scale questionnaire regarding physical and functional cutaneous signs to score from 0 to 10.
Soothing efficacy by a questionnaire | Change from just after application to 1 week and to 3 weeks later
  Subjects evaluate the soothing effect of the investigational product with a questionnaire
Cosmetic acceptability and efficacy perceived questionnaire | After 3 weeks of tested product
  Questionnaire with open questions and scales ranging from 0 to 10 where 0 was the worst satisfaction and 10 the best one.

CONTACTS AND LOCATIONS:
Overall Officials: Lexi LIU, Study Chair — EUROFINS CHINA
Locations (1):
- Eurofins China, Guangzhou, Haizhu District, China